CLINICAL TRIAL: NCT01440296
Title: Magnetic Resonance Imaging (MRI) Characterization of Carotid Plaque and Prediction of End-organ and Clinical Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Alan Moody, Dr, Sunnybrook Health Sciences Centre
Other Study IDs: CAIN-001
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Atherosclerosis; Carotid Artery Disease
MeSH Terms: conditions — Atherosclerosis; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The Canadian Atherosclerosis Imaging Network (CAIN) is a pan-canadian imaging network funded through grants from the Canadian Foundation for Innovation (CFI) and the Canadian Institutes of Health Research (CIHR). This unique research network is focused on the pathobiology of atherosclerotic disease as it pertains to the coronary and carotid circulations. The CAIN research program involves the creation of a unique national network focused on in vivo imaging of vessel wall disease, combined with imaging of occult end-organ disease as well as the acquisition of clinical and pathological end points. CAIN enables unprecedented cross-sectional and longitudinal clinical studies of patients with atherosclerotic disease in coronary or carotid vascular beds, and has established an international resource for studying the natural history, progression, regression and novel therapeutic interventions aimed at atherosclerosis.

The primary outcome of this study is to accurately characterise carotid plaque morphology in non-surgical patients with mild to severe (30-95%) carotid disease. The investigators will also assess evidence of ischaemic brain disease. Patients will undergo MRI scanning of the brain and carotid and US scanning of the carotid at baseline and thereafter at 1 and 2 years or sooner if presenting clinically in order to monitor the natural history of carotid atherosclerosis and its effect on end-organ brain disease.

Patients will consent to baseline scanning and follow up at 1 and 2 years, and databasing of clinical and imaging data. After each imaging session images will be processed, stored locally and also sent to a central repository. 500 patients will be recruited over a 2 year period in anticipation of study completion within 4 years.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients over the age of 18 years.
* written informed consent (approved by the Institutional Review Board [IRB]/Independent Ethics Committee [IEC]) obtained prior to any study specific procedures.
* patient with mild to severe carotid artery disease

Exclusion Criteria:

* any condition that would contra-indicate Magnetic Resonance Imaging or administration of contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients from tertiary care centre
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-03

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada